CLINICAL TRIAL: NCT00312780
Title: A Randomized, Double-Blind, Placebo-Controlled Study of XL784 Administered Orally to Subjects With Albuminuria Due to Diabetic Nephropathy
Brief Title: Study of XL784 in Patients With Albuminuria Due to Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL784-201
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Albuminuria; Diabetic Nephropathy
Keywords: albuminuria; diabetic nephropathy; diabetes
MeSH Terms: conditions — Albuminuria; Diabetic Nephropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: XL784 (Experimental)
  Interventions: Drug: XL784
- Arm 2: Placebo Gel capsules (Placebo Comparator)
  Interventions: Drug: XL784

INTERVENTIONS:
Drug: XL784 — XL784 softgel capsules (100 mg per capsule) orally administered at a dose of 200 mg/day (or placebo softgel capsules)

SUMMARY:
This clinical study is being conducted at multiple sites to determine the activity, safety and tolerability of XL784 when given daily to patients with albuminuria due to diabetic nephropathy. XL784 is a small molecule reno-protective metalloproteinase inhibitor, inhibiting both ADAMs (including ADAM10, a target of significant interest because of its important role in blood vessel formation and cell proliferation, and ADAM17/TACE, activation of which has been associated with renal deterioration) and MMPs (including MMP-2 and MMP-9). XL784 was specifically optimized to be MMP-1 sparing, which may be clinically significant because inhibition of MMP-1 has been hypothesized to be associated with musculoskeletal toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus with albuminuria, observed within 3 months of screening
* Prior to randomization, subject has a glomerular filtration rate (GFR) >/= 40 mL/min
* Prior to randomization, the subject has albuminuria defined as ACR >/= 500 mg/g
* Stable seated blood pressure at the screening visit and prior to randomization
* Subject has been on a stable dose and schedule of an angiotension converting enzyme (ACE) inhibitor and/or an angiotension receptor blocker (ARB) for at least 3 months before first dose of study drug
* If on antidiabetic medication, subject has been on a stable dose and schedule for at least 3 months prior to first dose of study drug
* Sexually active subjects must use an accepted method of contraception during the course of the study and for 3 months after
* Signed informed consent

Exclusion Criteria:

* Subject has participated in an investigational study and received an investigational drug within 30 days of the first dose of XL784
* Hemoglobin A1c (HbA1c) value of >10% at screening
* Subject has had either organ transplantation or is currently on immunosuppressive therapy
* Non-steroidal anti-inflammatory drugs (NSAIDs) within 5 days of urine screening assessments
* Current diagnosis of one or more of the following conditions: 1) infection requiring parenteral antibiotics, 2) urinary tract infection, 3) hepatic dysfunction or disease, 4) symptomatic congestive heart failure, 5) unstable angina pectoris, 5) serious cardiac arrhythmia
* Clinically evident diabetic gastroparesis or motility disturbance
* Proteinuria not due to diabetic nephropathy
* Diltiazem or verapamil
* Ongoing condition where treatment with NSAIDs is anticipated (aspirin </= 325 mg/day is allowed)
* Recent history of drug or alcohol abuse
* Pregnant or breastfeeding female subjects
* Known HIV and/or receiving anti-retroviral therapy
* Known allergy or hypersensitivity to any component of XL784 formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction in albumin excretion relative to creatinine | 27 weeks

SECONDARY OUTCOMES:
Safety and tolerability | 27 weeks
Pharmacokinetics and renal elimination | 27 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Aggarwal, MD, MBA, Study Director — Exelixis
Locations (45):
- United States (45):
  - Parkway Medical Center, Birmingham, Alabama
  - Winston Technology, Inc., Haleyville, Alabama
  - Redpoint Research, Phoenix, Arizona
  - International Clinical Research Network, Inc., Chula Vista, California
  - Scripps Clinic, Torrey Pines, Division of Nephrology, La Jolla, California
  - National Research Institute, Los Angeles, California
  - West Los Angeles VA Medical Center, Los Angeles, California
  - UCLA Medical Center, Center for the Health Sciences, Los Angeles, California
  - Arroyo Research Inc., Pasadena, California
  - Western Nephrology and Metabolic Bone Disease, PC, Lakewood, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC, Thornton, Colorado
  - Soundview Research Associates, Norwalk, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - MedStar Clinical Research Center, Washington D.C., District of Columbia
  - Clinical Research of South Florida, Coral Gables, Florida
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - Renal Associate of Baton Rouge, Baton Rouge, Louisiana
  - Intermed, Portland, Maine
  - MODEL Clinical Research, Baltimore, Maryland
  - Renal Unit, Joslin Diabetes Center, Boston, Massachusetts
  - Fallon Clinic Inc. at Worcester Medical Center, Department of Nephrology, Worchester, Massachusetts
  - Center for Urban and African American Health, Detroit, Michigan
  - South Mississippi Nephrology, Gulfport, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Creighton Dibetes Center, Omaha, Nebraska
  - University of Nebraska Medical Center - Nephrology, Omaha, Nebraska
  - LAND Clinical Studies, LLC, West Caldwell, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke South, Durham, North Carolina
  - Division of Nephrology/Department of Medicine, Case Western Rserve University, MetroHealth Medical Center Campus, Cleveland, Ohio
  - The Ohio State University Medical Center, Division of Nephrology, Columbus, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Nephrology Associates, PC, Nashville, Tennessee
  - Heartland Medical, PC, New Tazewell, Tennessee
  - Diabetes Center of the Southwest, Midland, Texas
  - dgd Research, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Health System, Nephrology Division, Charlottesville, Virginia
  - Zablocki Veterans Affairs Medical Center, Nephrology Section, Milwaukee, Wisconsin